CLINICAL TRIAL: NCT04111887
Title: Depression Prevention Programs: A Pilot Trial
Brief Title: Pilot Study Comparing Two Versions of Group Cognitive-behavioral Indicated Prevention Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Change Ahead
Record Dates: First submitted 2019-08-26; First posted 2019-10-01 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Change Ahead (Experimental): Each of the 6 weekly 1-hour sessions begins with a voluntary commitment to actively participate and to try something new in the upcoming week; includes a section devoted to selecting and publicly committing to one change focused on reducing negative/increasing positive cognitions and one change focused on increasing pleasant activities; and ends with home practice assignments. Additional exercises designed to increase dissonance induction include (a) group discussions for changing conditions, (b) roleplays to generate quick comebacks to written negative thoughts provided by other group members, (c) in-session writing exercises on the benefits of doing fun activities, (d) discussion of methods for creating internal and external accountability for positive change, (e) home practice assignment of engaging in actions to help someone else' mood, (f) writing a letter to my future self about positive intentions, and (g) providing positive feedback to other group members at the last session.
  Interventions: Behavioral: Group-based therapy
- Blues Program (Active Comparator): The 6 weekly 1-hour sessions begin with a review of concepts and (after Session 1) review of past home practice assignments; all sessions conclude with home practice assignments. Each session has a portion devoted to thought identification/recording and cognitive restructuring and a portion devoted to increased involvement in pleasant activities. We use motivational enhancement exercises to maximize willingness to use the new skills, behavioral techniques to reinforce use of the new skills, and group activities to foster feelings of group cohesion.
  Interventions: Behavioral: Group-based therapy
- Brochure control (Placebo Comparator): NIMH brochure that describes major depression and recommends treatment for depressed youth ("Let's Talk About Depression" NIH Pub. 01-4162), as well as information about local treatment options.
  Interventions: Behavioral: Group-based therapy

INTERVENTIONS:
Behavioral: Group-based therapy — College students with depressive symptoms will be randomized to one of three conditions: 1) a cognitive behavioral prevention intervention, 2) a cognitive behavioral prevention intervention with counter-attitudinal elements or 3) an educational brochure control. We will test if the additional of counter attitudinal elements produces intervention effects when delivered to participants with sub threshold depressive symptoms.

SUMMARY:
The purpose of this study is to compare the effectiveness of two depression prevention programs and a control brochure for college students. Participants may experience reductions in depressive symptoms and prevention of future depression.

ELIGIBILITY:
Inclusion Criteria:

* current student at the University of Oregon
* subthreshold symptoms of depression, as indicated by a CES-D depression screener score of 20 or greater

Exclusion Criteria:

* current diagnosis of major depression
* acute suicidal ideation requiring immediate mental health treatment

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline Depressive Disorder Diagnostic using the Kiddie Schedule for Affective Disorders and Schizophrenia at 6 weeks, 3 months and 6 months | Measured at baseline, 6 weeks, 3 months and 6 months
  Evaluate change (if any) by using the Kiddie Schedule for Affective Disorders and Schizophrenia at the 6 week, 3 month and 6 month marks.
Difference in attendance in Change Ahead vs Blues Program groups using group leader notes | Measured at each group therapy session (6 weeks in total).
  Evaluate difference (if any) in attendance in Change Ahead vs Blues Program group therapies by using group leader notes.
Difference in future onset of Major Depressive Disorder using the Kiddie Schedule for Affective Disorders and Schizophrenia | Measured at baseline, 6 weeks, 3 months and 6 months.
  Evaluate difference (if any) in the future onset of Major Depressive Disorder at 3 months and 6 months.

SECONDARY OUTCOMES:
Activity level | Measured at baseline, weeks 2,4 and 6.
  Evaluate the participants activity levels using Ecological Momentary Assessments (EMAs).
Emotions | Measured at baseline, weeks 2,4 and 6.
  Evaluate the participants emotions using Ecological Momentary Assessments (EMAs).
Positive and negative thoughts | Measured at baseline, weeks 2,4 and 6.
  Evaluate the participants positive and negative thoughts using Ecological Momentary Assessments (EMAs).
Assessments using writing samples | Measured at baseline and 6 weeks
  Evaluate difference (if any) in social and academic problem solving skills and thoughts of the future.
Depression and anxiety symptoms using the PHQ-9 | Measured at baseline, 6 weeks, 3 months and 6 months
  Evaluate difference (if any) in self-reported depression and anxiety symptoms
Depression and anxiety symptoms using the GAD-7 | Measured at baseline, 6 weeks, 3 months and 6 months
  Evaluate difference (if any) in self-reported depression and anxiety symptoms
Social adjustment in school, work, peer, spare time, and family domains | Measured at baseline, 6 weeks, 3 months and 6 months
  Evaluate difference (if any) in self-reported social adjustment using 17 items adapted from Social Adjustment Scale-Self Report for Youth (Weissman, Orvaschel, & Padian, 1980)
Negative life events | Measured at baseline
  Evaluate difference (if any) in self-reported negative life events
Health care utilization | Measured at baseline, 6 weeks, 3 months and 6 months
  Evaluate difference (if any) in self-reported utilization of health care services for physical health problems/injuries, mental health problems, and other personal problems.
Negative automatic thoughts | Measured at baseline, 6 weeks, 3 months and 6 months
  Evaluate difference (if any) in self-reported negative automatic cognition using 12 items from the Automatic Thoughts Questionnaire (ATQ; Hollon & Kendall, 1980)
Negative attributional style | Measured at baseline, 6 weeks, 3 months and 6 months
  Evaluate difference (if any) in self-reported negative attributional style
Substance use | Measured at baseline (in intake screener), 6 weeks, 3 months and 6 months
  Evaluate difference (in any) in self-reported substance use using 10 items from Stice, Barrera and Chassin (1998). Participants report the frequency of intake of beer/wine/wine coolers and hard liquor, frequency of heavy drinking (5 or more drinks in a row), frequency of times drunk, and frequency of marijuana, stimulants, downers, inhalants, and hallucinogen use.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States